CLINICAL TRIAL: NCT06578559
Title: Single Arm Phase II Study of ctDNA-guided Encorafenib Plus Cetuximab Retreatment in Patients With BRAF V600E Mutated mCRC (BRICKET)
Brief Title: Phase II Study of ctDNA-guided Encorafenib Plus Cetuximab Retreatment in Patients BRAF V600E Mutated mCRC
Acronym: BRICKET
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRICKET
Record Dates: First submitted 2024-07-29; First posted 2024-08-29 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
Keywords: ctDNA; Encorafenib; Cetuximab; rechallenge; retreatment; BRAF V600E
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Encorafenib + Cetuximab (Experimental)
  Interventions: Drug: Cetuximab; Drug: Encorafenib

INTERVENTIONS:
Drug: Cetuximab — 500 mg/sqm intravenous infusion over 120-minute at cycle 1 (if well tolerated, it is administered over 90 minutes at second administration, and over 60 minutes by the third administration) every 14 days.
Drug: Encorafenib — 300 mg once daily (four 75 mg oral capsules).

SUMMARY:
The aim of this study is to evaluate the activity, in terms of best response according to RECIST criteria 1.1 as assessed by the local investigator, of the ctDNA-guided retreatment with encorafenib plus cetuximab in BRAFV600E mutated mCRC patients experiencing benefit from previous exposure to encorafenib plus cetuximab (+/- chemotherapy) and with BRAFV600E mutated, KRAS, NRAS and MAP2K1 wild-type and MET not amplified status on ctDNA at the time of study entry.

DETAILED DESCRIPTION:
This is a proof-of-concept, multicenter, open-label, single arm one-stage phase II trial of a ctDNA-guided retreatment with encorafenib plus cetuximab for mCRC patients bearing the BRAFV600E mutation and with the key following characteristics:

* initial benefit and then secondary resistance to a previous exposure to encorafenib and cetuximab with or without chemotherapy;
* only one subsequent intervening anti-BRAF and anti-EGFR-free line of therapy;
* confirmed BRAFV600E mutated status and no detectable mutations in KRAS, NRAS, MAP2K1 and no amplification of MET in ctDNA at the time of retreatment;

Eligible patients will receive Encorafenib 300 mg once daily (four 75 mg oral capsules) and Cetuximab 500 mg/sqm iv infusion every 14 days.Treatment will be delivered in 28-day cycles until disease progression, unacceptable toxic effects, withdrawal of consent, initiation of subsequent anticancer therapy, or death.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven diagnosis of colorectal adenocarcinoma;
* age ≥ 18 years;
* ECOG Performance status ≤ 1;
* BRAFV600E mutated status of primary colorectal cancer and/or related metastasis, by local laboratory assessment according to standard procedures by means of molecular assay on genomic DNA;
* Metastatic disease with at least one measurable lesion according to RECIST 1.1. criteria;
* previous treatment with encorafenib plus cetuximab with or without chemotherapy (i.e., ±FOLFOX/FOLFIRI) in any line, producing a RECIST 1.1 complete/partial response or disease stabilisation, with a PFS of this treatment lasting at least 6 months;
* documentation of RECIST 1.1 disease progression during or after the end of the previous exposure to encorafenib plus cetuximab ± chemotherapy;
* one intervening line of treatment not including any BRAF and EGFR inhibitor, between the end of first exposure to encorafenib plus cetuximab ± chemotherapy and the time of screening;
* at least 4 months elapsed between the end of the previous exposure to encorafenib plus cetuximab ± chemotherapy and the retreatment with encorafenib plus cetuximab;
* previous treatment with immune checkpoint inhibitors (anti-PD-1/PD-L1 alone or in combination with anti-CTLA-4 agent), in the case of MSI-H or dMMR mCRC;
* availability of blood sample for ctDNA analysis within 28 days prior enrolment;
* BRAFV600E mutated status of ctDNA at screening (central laboratory assessment by means of GUARDANT360 CDx, Guardant Health);
* KRAS, NRAS, MAP2K1 wild-type status and MET not amplified status in ctDNA at screening (central laboratory assessment by means of GUARDANT360 CDx, Guardant Health);
* Availability of archival tumour tissue (primary tumour and/or metastases) for biomarker analysis;
* neutrophils >1.5 x 109/L, Platelets >100 x 109/L, Hgb >9 g/dl. Transfusions will be permitted provided the patient has not received more than two units red blood cells in the prior 4 weeks to achieve this criterion.
* adequate renal function characterised by serum creatinine ≤ 1.5 × upper limit of normal (ULN), or calculated by Cockroft-Gault formula or directly measured creatinine clearance ≥ 50 mL/min at screening;
* adequate hepatic function characterised by the following at screening: Serum total bilirubin ≤ 1.5 × ULN and < 2 mg/dL. Note: Patients who have a total bilirubin level > 1.5 × ULN will be allowed if their indirect bilirubin level is ≤ 1.5 × ULN; Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 × ULN, or ≤ 5 × ULN in presence of liver metastases. In the presence of documented Gilbert's syndrome, a value of total bilirubin < 3 × ULN is acceptable.
* adequate electrolytes at baseline, defined as serum potassium and magnesium levels within institutional normal limits (Note: replacement treatment to achieve adequate electrolytes will be allowed).
* INR or aPTT ≤ 1.5 × ULN;
* QT interval corrected for heart rate ≤480 msec at screening;
* ability to take oral medications;
* women of childbearing potential must have a negative blood pregnancy test at the screening. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least twelve continuous months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;
* subjects and their partners must be willing to avoid pregnancy from the study screening until 1 month after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator. Encorafenib may decrease the efficacy of hormonal contraceptives. Therefore, female patients using hormonal contraception are advised to use an additional or alternative method such as a barrier method (i.e., condom) from the screening phase for at least 1 month following the last dose of study treatment. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;
* written informed consent to study procedures;
* life expectancy of at least twelve weeks;
* will and ability to comply with the protocol.

Exclusion Criteria:

* Known hypersensitivity or contraindications to trial drugs or any component of the trial drugs;
* discontinuation of previous treatment with encorafenib and/or cetuximab with or without chemotherapy due to encorafenib- and/or cetuximab-related adverse events;
* symptomatic brain metastases or spinal cord compression. Notes: Patients previously treated or untreated for these conditions who are asymptomatic in the absence of corticosteroid and anti-epileptic therapy are allowed. Brain metastases or spinal cord compression must be stable for ≥ 4 weeks, with imaging (e.g., magnetic resonance imaging [MRI] or computed tomography [CT]) demonstrating no current evidence of progressive brain metastases or spinal cord compression at screening;
* leptomeningeal disease;
* other co-existing malignancies or malignancies diagnosed within the last 5 years except for adequately treated localised basal and squamous cell carcinoma or cervical cancer in situ;
* treatment with any investigational drug within 30 days prior to enrolment or two investigational agent half-lives (whichever is longer);
* Impaired gastrointestinal function (i.e., uncontrolled nausea, vomiting or diarrhea, malabsorption syndrome, small bowel resection) or disease which may significantly alter the absorption of oral study intervention or recent changes in bowel function suggesting current or impending bowel obstruction;
* use of any herbal medications/supplements or any medications or foods that are moderate or strong inhibitors or inducers of CYP3A4/5 ≤1 week prior to the start of treatment;
* diagnosis of interstitial pneumonitis or pulmonary fibrosis;
* known history of acute or chronic pancreatitis within 6 months prior to the start of the treatment;
* history of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention immunomodulatory or immunosuppressive medications or surgery) ≤12 months prior to first dose;
* impaired hepatic function, defined as Child-Pugh class B or C;
* clinically significant cardiovascular diseases, including any of the following:

  * history of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft, coronary angioplasty or stenting) ≤6 months prior to registration;
  * congestive heart failure requiring treatment (New York Heart Association Class II and above);
  * recent history (within 1 year prior to registration) or presence of clinically significant cardiac arrhythmias (including uncontrolled atrial fibrillation or uncontrolled paroxysmal supraventricular tachycardia);
* QT interval corrected for heart rate >480 msec at screening and rate uncontrolled atrial fibrillation and paroxysmal supraventricular tachycardia;
* pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barrier contraceptive measure or oral contraception) from the screening phase until 1 month after the last trial treatment;
* residual CTCAE ≥ Grade 2 toxicity from any prior anticancer therapy, with the exception of grade 2 alopecia or grade 2 neuropathy
* active eye disorders, including keratitis, ulcerative keratitis or severe dry eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 8 months after the enrollment of the last patient.
  The percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria. The determination of clinical response will be based on investigator-reported measurements.
  Responses will be evaluated with a total body computed tomography (CT) scan every 8 weeks.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 8 months after the enrollment of the last patient.
  The time interval computed from the date of study enrollment to the date of objective progression according to the RECIST criteria (version 1.1) or death, whatever comes first.
  Patients alive and free of progression prior to the analysis cut-off date are censored at the date of the last disease assessment.
Overall Survival (OS) | 8 months after the enrollment of the last patient.
  The time from the date of study enrollment to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Overall Toxicity Rate | 8 months after the enrollment of the last patient.
  The percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (CTCAE version 5.0).
  The CTCAE are classified as Grades 1 to 5 (from milder to more severe symptoms).
Grade 3/4 Toxicity Rate | 8 months after the enrollment of the last patient.
  The percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (CTCAE version 5.0).
  The CTCAE are classified as Grades 1 to 5 (from milder to more severe symptoms).
Early Objective Response Rate (EORR) | 8 months after the enrollment of the last patient.
  The percentage of patients, relative to the total of the enrolled subjects, achieving at least a 20% decrease in the sum of diameters of RECIST target lesions at week 8 compared to baseline.
Depth of Response (DpR) | 8 months after the enrollment of the last patient.
  The relative change in the sum of longest diameters of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline.
Objective Response Rate in the screening failure population (ORR-failure) | 8 months after the enrollment of the last patient.
  Best objective response according to RECIST 1.1 criteria of the first line after ctDNA screening failure, if administered.
Progression Free Survival in the screening failure population (PFS-failure) | 8 months after the enrollment of the last patient.
  The time interval computed from the start of the first treatment after ctDNA screening failure, if delivered, to the date of objective progression according to the RECIST criteria (version 1.1) or death, whichever comes first.
Overall Survival in the screening failure population (OS-failure) | 8 months after the enrollment of the last patient.
  The time interval computed from the start of the first treatment after ctDNA screening failure, if delivered, to the date of death due to any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). | Questionnaires will be administered at baseline (cycle 1 day 1), every 8 weeks thereafter, at disease progression and after 30 days following end of study treatment.
  The EORTC QLQ-C30 contains functional scales, symptom scales, single items scale and a global health status/QoL scale. Raw scores are standardized and converted into scale scores ranging from 0 to 100.
  Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
  Quality of life will be evaluated for patients who will have completed at least one questionnaire item at baseline and during the study period through descriptive summary statistics.
Quality of Life as assessed by the European Organization for Research and Treatment of Cancer Quality of Life Module for Colorectal cancer 29 (EORTC QLQ-CR29). | Questionnaires will be administered at baseline (cycle 1 day 1), every 8 weeks thereafter, at disease progression and after 30 days following end of study treatment.
  The EORTC QLQ-CR29 includes 29 items that evaluate symptoms (gastrointestinal, urinary, pain and others) and functional areas (sexual, body image and others) that are associated with CRC and its treatments.
  There are separate items for patients with and without a stoma and separate items to evaluate the sexual function of men and women. Raw scores are standardized and converted into scale scores ranging from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms on the symptom scales.
  Quality of life will be evaluated for patients who will have completed at least one questionnaire item at baseline and during the study period through descriptive summary statistics.
Time To Deterioration in Quality of Life (TTD) | 8 months after the enrollment of the last patient.
  The time from baseline to the first onset of a 10-point or greater decrease from study enrollment for functional scales or a 10-point or greater increase for symptom scales or death.

CONTACTS AND LOCATIONS:
Overall Officials: Carlotta Antoniotti, MD, PhD, Principal Investigator — Department of Translational Research and New Technologies in Medicine and Surgery - University of Pisa
Locations (13):
- Italy (13):
  - L'Azienda Ospedaliero Universitaria di Cagliari, Monserrato, CA
  - Istituto Romagnolo Per Lo Studio Dei Tumori "Dino Amadori" Irccs Irst, Meldola, FC
  - Fondazione Casa Sollievo Della Sofferenza - Irccs, San Giovanni Rotondo, FG
  - Pia Fondazione di Culto e di Religione Cardinale G. Panico, Tricase, LE
  - IRCCS Istituto Nazionale dei Tumori di Milano, Milan, MI
  - Istituto Oncologico Veneto Irccs, Padua, PD
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, PI
  - Nuovo Ospedale di Prato S. STEFANO, Prato, PO
  - AUSL Romagna, Ravenna, RA
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - A.O.U. Citta Della Salute E Della Scienza Di Torino Presidio Molinette, Turin, TO
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine, UD
  - Azienda Ospedaliera Universitaria degli Studi di Campania L. Vanvitelli, Naples

IPD SHARING:
Plan to Share IPD: No